CLINICAL TRIAL: NCT05491148
Title: Study of the Functional State of the Body of Medical Workers in the Intensive Care Unit for Newborns
Status: Completed | Type: Observational
Sponsor: Federal State Budgetary Scientific Institution "Izmerov Research Institute of Occupational Health" (Other)
Responsible Party: Principal Investigator, Andrey Mikhailovich Geregey, Head of the Laboratory of Personal Protective Equipment and Industrial Exoskeletons Andrey Geregey, Federal State Budgetary Scientific Institution "Izmerov Research Institute of Occupational Health"
Other Study IDs: PPE-06
Record Dates: First submitted 2022-08-04; First posted 2022-08-08 (Actual); Last update posted 2023-05-16 (Actual); Status verified 2023-05

CONDITIONS: Сhanges in the Cardiovascular System in Healthcare Workers During Work Shift
Keywords: functional state of the body; medical personnel; heart rate variability; cognitive functions; cardiovascular system
MeSH Terms: interventions — Working Conditions

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- medical workers: medical workers of the resuscitation and intensive care unit of newborns
  Interventions: Other: work conditions

INTERVENTIONS:
Other: work conditions — an increased degree of responsibility for the life of newborns, high psycho-emotional stress, intellectual stress, an irrational work and rest regime, in connection with the COVID-19 pandemic, also using personal protective equipment against biological factors

SUMMARY:
The purpose of this work is to assess the functional state of the body of medical workers in the neonatal resuscitation and intensive care unit in the conditions of work.

ELIGIBILITY:
Inclusion Criteria:

* the volunteer has practical experience in the neonatal intensive care unit
* digestive tract, kidney, cardiorespiratory system, mervous system or musculoskeletal system pathology

Exclusion Criteria:

* acute and chronic diseases of the cardiovascular, bronchopulmonary, neuroendocrine systems, musculoskeletal system, as well as diseases of the gastrointestinal tract, liver, kidneys
* body temperature above 37 ° C, heart rate over 90 beats / min, systolic and diastolic blood pressure above 140 mm Hg. Art. and 90 mm Hg. Art.
* organic brain lesions, increased convulsive activity in history
* receiving more than 10 units. alcohol per week or history of alcoholism, drug addiction, drug abuse

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Healthy medical workers in neonatal intensive care unit
Sampling Method: Probability Sample
Enrollment: 17 (Actual)
Dates: Start 2022-08-29 (Actual); Primary Completion 2022-10-05 (Actual); Study Completion 2022-10-10 (Actual)

PRIMARY OUTCOMES:
Heart rate | 8 hours
  bpm, "Armed": "YE-630A" (ТМ "ARMED", Russia)
Blood pressure | 8 hours
  mm Hg, "Armed": "YE-630A" (ТМ "ARMED", Russia)
Anthropometry (Height) | 1 hour
  Height (cm), weight (kg), Seca 703 ("Seca GMBH&Co", Germany)
Anthropometry (Weight) | 1 hour
  Weight (kg), Seca 703 ("Seca GMBH&Co", Germany)
Body temperature | 1 hour
  Celsius, Thermoval Standard ("PAUL HARTMANN", Germany)
Electrocardiography | 1 hour
  Electrocardiogram analysis, Electrocardiographic system "Poly-Specter-SM" (LLC "Neurosoft", Russia)
Cognitive functions test 1 | 1 hour
  Bourdon correction test, Universal psychodiagnostic complex NS-Psychotest (LLC "Neurosoft", Russia)
Cognitive functions test 2 | 1 hour
  Simple visual-motor reaction test, Universal psychodiagnostic complex NS-Psychotest (LLC "Neurosoft", Russia)
Cognitive functions test 3 | 1 hour
  Growing account test. Universal psychodiagnostic complex NS-Psychotest (LLC "Neurosoft", Russia)

SECONDARY OUTCOMES:
Survey | 1 hour
  Subjective survey on functional state of the body (7 scales)

CONTACTS AND LOCATIONS:
Overall Officials: Inga Malakhova, Principal Investigator — Junior scientist
Locations (1):
- Federal State Budgetary Scientific Institution Izmerov Research Institute of Occupational Health, Moscow, Russia

IPD SHARING:
Plan to Share IPD: No